CLINICAL TRIAL: NCT04993131
Title: Liver Transplantation for Non-resectable Perihilar Cholangiocarcinoma: a Prospective Exploratory Trial
Brief Title: Liver Transplantation for Non-resectable Perihilar Cholangiocarcinoma
Acronym: TESLA II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Sheraz Yaqub, Assoc Professor, MD PhD FEBS, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 270331
Record Dates: First submitted 2021-07-02; First posted 2021-08-06 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Perihilar Cholangiocarcinoma; Klatskin Tumor; Bile Duct Cancer
MeSH Terms: conditions — Klatskin Tumor; Bile Duct Neoplasms | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liver transplant (Experimental): The patients will be transplanted according to standard procedures by the institutional protocol. Median time of surgery is 7 hours and 20 minutes. Each surgical procedure will be performed by specialists at the Rikshospitalet liver transplantation team, which consists of seven specialists at the unit. The transplantation procedure is initiated by an exploratory laparotomy with clinical assessment and frozen section of the lymphnodes in the hepatoduodenal ligament and along the common hepatic artery/coeliac axis. Complete clearance of the lymphatic tissue around the hepatoduodenal ligament. Frozen section is obtained from the distal end of the common bile duct. Evidence of disease dissemination to these regional lymph nodes will be an absolute contraindication to transplantation.
  Interventions: Procedure: Liver transplant

INTERVENTIONS:
Procedure: Liver transplant — Liver transplant.

SUMMARY:
The study will investigate whether liver transplantation provides increased survival, low side effects and good quality of life in patients with bile duct cancer where the tumor cannot be removed by normal surgery. Analyzes of blood and tissue samples from the tumor will be investigated to see if the analyzes can indicate who may have recurrence of the disease after liver transplantation. Furthermore, the effect of chemotherapy on normal liver and tumor tissues in the liver that are removed during transplantation will be investigated.

DETAILED DESCRIPTION:
Liver transplantation (Lt) is an established method of treatment for acute and chronic liver failure. One and five- year survival after Lt is approximately 90% and 80%, respectively. Currently, Lt is a treatment option for selected patients with primary carcinomas in the liver and in patients with liver metastases from neuroendocrine tumors. The prerequisite is that there is no extra-hepatic tumor growth and that the primary tumor is removed. Lt for cancer comprises of 14% of all Lts in Europe (www.etlr.org). Types of primary carcinomas eligible for transplantation today include hepatocellular carcinoma (HCC), hepatoblastoma, hemangioendothelioma, and perihilar cholangiocarcinoma (pCCA), the latter in clinical protocols. The most common secondary hepatocarcinomas are neuroendocrine tumours (carcinoid tumours and gastrinomas). The International Registry of Hepatic Tumors in Liver Transplantation show that survival of HCC patients after transplantation is above 70% and 60% at 1 and 5 years, respectively. Recent studies on HCC and liver transplantation have shown even better results when patients are treated with an immunosuppressive regimen containing the antiproliferative agent rapamycin. For hepatoblastoma (children) and malign hemangioendotheliaoma the five-year survival is between 50-60% and for intestinal sarcomas and neuroendocrine tumours it is approximately 35-40%. In patients transplanted for pCCA using a multimodal approach utilizing neoadjuvant radiation, chemotherapy and liver transplantation (Mayo protocol) 5-year patient survival of >80% in selected patients compared to a corresponding 21% five-year survival in liver resection.

Malignancy of the biliary tree (cholangiocarcinoma, CCA) is a rare cancer with an annual incidence around 150 cases in Norway. Cholangiocarcinoma can be subdivided into distal, perihilar, and intrahepatic according to their anatomical location5. Although rare, intrahepatic cholangiocarcinoma (iCCA) constitutes the second most common primary liver cancer after hepatocellular carcinoma, and the worldwide incidence of iCCA is increasing. Despite improvements in multidisciplinary management, patients with CCA have a poor outcome and only 20% of patients are eligible for surgical resection, with 5-year overall survival of less than 10% for all patients. The only potentially curative treatment option is surgical resection with complete excision of tumor with negative margins.

An Irish study with liver transplantation for patients with unresectable hilar CCA who received neoadjuvant chemoradiotherapy had 1- , 3- and 5-year survival of 81%, 69% and 62% respectively, of the transplanted patients. We have recently started a prospective exploratory study, TESLA trial, investigating Lt in non-resectable iCCA with stable disease on oncological treatment.

Building on these results in addition to our own experience with liver transplantation for non-resectable colorectal liver metastases, we want to investigate in the TESLA-II trial the role of Lt in selected patients with unresectable pCCA, who fulfill the inclusion criteria.

ELIGIBILITY:
Inclusion criteria

* Radiologically strong suspicion of pCCA
* Tumor can involve intrahepatic portal vein without thrombosis of extrahepatic portal vein
* Tumor can involve hepatic artery distal to gastroduodenal artery or involve replaced hepatic artery
* First time pCCA
* Disease deemed not eligible for liver resection based on tumor location or underlying liver dysfunction
* No extrahepatic disease, or lymph node involvement detected on imaging
* No signs of extrahepatic metastatic disease according to PET-CT scan
* No signs of extrahepatic metastatic disease according to CT or MR (chest/abdomen/pelvis) scan within 4 weeks prior to the faculty meeting at the transplant unit
* At least 18 years of age
* Good performance status, Eastern Cooperative Oncology Group (ECOG) score: 0 or 1
* Satisfactory blood tests Hb >10g/dl, neutrophiles >1.0 (after any G-CSF), TRC >50, Bilirubin<3 x upper normal level, ASAT, ALAT<5 x upper normal level, Creatinine <1.5 x upper normal level. Albumin above lower normal level, Normal IgG4 levels
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to GCP, and national/local regulations
* Received chemotherapy for at least 6 months with at least 10% response according ti RECIST criteria and with no progression of disease at time of Lt
* At least 10 months from diagnosis
* Patient must be accepted for transplantation before progressive disease
* Twelve months or more time span from the diagnosis of pCCA and date of being listed for liver transplantation

Exclusion criteria

* Tumor involving common hepatic artery, celiac trunck or superior mesenteric artery the tumor
* Tumor involving main portal vein
* Tumor involving inferior vena cava
* Perforation of the visceral peritoneum
* Weight loss >15% the last 6 months
* Patient BMI > 30
* Other malignancies, except curatively treated more than 5 years ago without relapse
* Known history of human immunodeficiency virus (HIV) infection
* Prior history of solid organ or bone marrow transplantation
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known hypersensitivity to rapamycin
* Prior extrahepatic metastatic disease
* Women who are pregnant or breast feeding
* Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2035-05-31 (Estimated); Study Completion 2045-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From screening and until 36 months after inclusion
  Patient record

SECONDARY OUTCOMES:
Overall survival from time of relapse | From time of relapse and until 36 months after inclusion
  Patient record
Disease free survival | After liver transplantation and up 10 years after liver transplantation
  CT-scan/MRI scan according to RECISTcriteria
Time to start of new treatment/change in strategy | Immediately after liver transplatation to start of new treatment
  Patient record
Quality of life (EORTC QLQ-C30), time to decrease in physical function and global health score | Up to 10 years after liver transplantation
  Quality of life measured by EORTC QLQ-C30
Complication according to Clavien-Dindo grad 3-5 | Up to 90 days after liver transplantation
  Patient record
Diagnosis of other malignancies | Up to 10 years after liver transplantation
  Patient record
Survival in relation to biological markers | After Liver Transplant until 10 years after liver transplantation
  CA19-9, CEA

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo university hospital, Oslo, Norway